CLINICAL TRIAL: NCT01725906
Title: Genotypic Resistance Guided Therapy in the Treatment of Helicobacter Pylori Infection
Brief Title: Genotypic Resistance Guided Therapy in Helicobacter Pylori Eradication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Doctor, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201202068MIC
Record Dates: First submitted 2012-10-31; First posted 2012-11-14 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Self Efficacy
Keywords: genotypic resistance guided therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Empirical therapy (Active Comparator): selection of antibiotic according to medication history
  Interventions: Drug: empirical therapy
- Genotypic resistance guided therapy (Experimental): selection of antibiotics according to genotypic resistance
  Interventions: Drug: Genotypic resistance guided therapy

INTERVENTIONS:
Drug: empirical therapy — 1. Nexium (esomeprazole), 40mg, bid, 14 days, plus
  2. Amoxicillin (Amoxicillin Trihydrate), 1gm, bid, 7 days, plus
  3. Flagyl (metronidazole), 500mg, bid, 7 days, plus either one of the following drugs
  4. Select either one of the drugs according to medication history Cravit (levofloxacin) , 250 mg, bid, D8-14 Klaricid (clarithromycin), 500 mg, bid , D8-14 Tetracycline, 500 mg, bid, D8-14
  Other Names: selection of antibiotics according to medication history
  Arms: Empirical therapy
Drug: Genotypic resistance guided therapy — 1. Nexium (esomeprazole), 40mg, bid, 14 days, plus
  2. Amoxicillin (Amoxicillin Trihydrate), 1gm, bid, 7 days, plus
  3. Flagyl (metronidazole), 500mg, bid, 7 days, plus either one of the following drugs
  4. Select either one of the drugs according to genotypic resistance results Cravit (levofloxacin) , 250 mg, bid, D8-14 Klaricid (clarithromycin), 500 mg, bid , D8-14 Tetracycline, 500 mg, bid, D8-14
  Other Names: selection of antibiotic according to genotypic resistance
  Arms: Genotypic resistance guided therapy

SUMMARY:
We aimed to compare the efficacy of genotypic resistance guided sequential therapy vs. empiric therapy in the third line therapy. Factors affecting the eradication rates, including the antibiotic resistance, CYP2C19 polymorphism, CagA and VacA status will also be assessed.

DETAILED DESCRIPTION:
The primary aim of this study is to compare the regimens selected using either one of the method (1) genotypic resistance guided versus (2) medication history guided therapy. (rather than to compare the efficacy of any drugs).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged greater than 20 years who have persistent H. pylori infection after at least two treatments and are willing to receive third line rescue regimens are considered eligible for enrollment.

Exclusion Criteria:

* Patients will be excluded from the study if any one of the following criteria is present: (1) children and teenagers aged less than 20 years, (2) history of gastrectomy, (3)gastric malignancy, including adenocarcinoma and lymphoma, (4) previous allergic reaction to antibiotics (Amoxicillin, Klaricid, Cravit) and prompt pump inhibitors (esomeprazole), (5)contraindication to treatment drugs, (6) pregnant or lactating women, (7) severe concurrent disease.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2012-11; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Eradication rate after third line rescue therapy | 8 weeks
  Primary End Point: Eradication rate will be evaluated according to Intent-to-treat (ITT) and per-protocol (PP) analyses.
  (genotypic resistance versus empirical therapy) Urea breath test will be used to determine the eradication status

SECONDARY OUTCOMES:
eradication rates in subgroup analysis by antibiotic resistance and regimen | 8 weeks
  eradication rate in subgroup analysis according to antibiotic resistance and treatment regimen

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Ming Liou, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan Universtiy Hospital, Taipei
  - National Taiwan University Hospital, Yun-Lin Branch, Yun-Lin County

REFERENCES:
- [Derived] Liou JM, Chen PY, Luo JC, Lee JY, Chen CC, Fang YJ, Yang TH, Chang CY, Bair MJ, Chen MJ, Hsu YC, Hsu WF, Chang CC, Lin JT, Shun CT, El-Omar EM, Wu MS; Taiwan Gastrointestinal Disease and Helicobacter Consortium. Efficacies of Genotypic Resistance-Guided vs Empirical Therapy for Refractory Helicobacter pylori Infection. Gastroenterology. 2018 Oct;155(4):1109-1119. doi: 10.1053/j.gastro.2018.06.047. Epub 2018 Jun 30. PMID 29964036